CLINICAL TRIAL: NCT05796817
Title: Reducing Oxygen Consumption in Critical Care (ROCC)
Brief Title: Reducing Oxygen Consumption in Critical Care
Acronym: ROCC
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 310355
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ventilator modification — The ventilator modification will be fitted to a ResMed Lumis 150, Breas® Nippy 4+ or Vivo 1, 2 or 3 ventilator. The participants oxygen level will be measured with and without the modification in place at their baseline ventilation, and with 1, 2 and 3 litres oxygen extra to their baseline. the researcher will then leave the modification on and slowly reduce the oxygen going into the ventilator, maintaining the participants SP02 at an acceptable level (>95%)

SUMMARY:
In normal practice oxygen supply can be easily met with existing hospital infrastructure. COVID - 19 however results in lung damage which greatly increases the amount of oxygen patients require - as a consequence some hospitals in the UK and other countries had situations where there was not enough oxygen for their inpatients.

COVID - 19 has caused many more patients to requiring assistance with their breathing using a ventilator. Due to the limited supply of sophisticated ventilators that 're-use' oxygen patients breathe out, some hospitals have used ventilators normally used by patients at home (domiciliary ventilators). Whilst these are inexpensive and commonly available, any oxygen the patient breathes out is simply released into the atmosphere.

The address this problem, and in turn reduce the oxygen demand on hospital infrastructure the biomedical engineering team (BME) at the Royal Brompton Hospital, London devised a simple 3-D printed modification which captures and reuses oxygen on commonly used domiciliary ventilators. Laboratory testing found this modification can increase the oxygen given by the ventilator without increasing the oxygen consumption of the ventilator - effectively reducing oxygen demand on hospital infrastructure.

This study will evaluate this modification in patients admitted to intensive care requiring assistance with their breathing. This will involve measuring oxygen levels on domiciliary ventilators (Breas Nippy 4+, ResMed Lumis 150 or Vivo 1, 2 or 3) with and without the modification and with small increases in oxygen supplied to the patient for a total study period of 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient in critical care using a ResMed LumisTM 150, Breas® Nippy 4+ or Vivo 1, 2 or 3 ventilator or deemed safe by treating consultant safe to switch to one.
* 28% or more of entrained oxygen (FiO2)
* Judged to be safe to tolerate increased fraction of inspired oxygen for periods of 10 minutes
* Arterial line insitu for clinical reasons

Exclusion Criteria:

* Thought to be clinically unstable during study protocol (2 hours)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients in critical care
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Arterial blood gas analysis - baseline | After 10 minutes
  PaO2 with and without modification fitted

SECONDARY OUTCOMES:
Arterial blood gas - modification and oxygen change | After 10 minutes of each experimental condition
  Oxygenation with and without modification in place with 1, 2 and 3 litres added to baseline FiO2
Arterial blood gas - CO2 | After 10 minutes of each experimental condition
  Arterial CO2 levels at each experimental condition

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Brompton and Harefield Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No